CLINICAL TRIAL: NCT00139243
Title: A Phase I/II Study of Taxotere, Cisplatin, 5-Fluorouracil and Leucovorin for Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Taxotere, Cisplatin, 5-Fluorouracil, and Leucovorin for Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sanofi (Industry); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-130
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Squamous Cell Carcinoma; Carcinoma of Head and/or Neck
Keywords: squamous cell carcinoma; Taxotere; carcinoma of head/neck; Cisplatin; 5-Fluorouracil; Leucovorin
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Docetaxel; Cisplatin; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Taxotere
Drug: Cisplatin
Drug: 5-Fluorouracil
Drug: Leucovorin

SUMMARY:
The purpose of this study is to determine the safety and maximum tolerated dose of the combination taxotere, cisplatin, 5-fluorouracil and leucovorin. We will also preliminarily assess whether the combination is effective in treating squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
* Patients will be premedicated at home with dexamethasone and leucovorin.
* On the first day of treatment, the patient will receive taxotere intravenously for one hour. Approximately one hour after the taxotere is completed, the patient will receive a 4 hour infusion of cisplatin and begin a four day continuous infusion of 5-fluorouracil and leucovorin. The infusion of 5-fluorouracil and leucovorin will be completed at home with the use of an infusion pump. This process will be repeated every 21-35 days (1 cycle) depending upon how quickly the patient recovers from the chemotherapy.
* During each cycle blood tests will be performed weekly. During the first cycle a physical exam will be performed weekly and then halfway through each subsequent cycle and immediately prior to the start of each subsequent cycle.
* At the end of each cycle the impact of the chemotherapy will be assessed. If after 2 cycles the cancer has not responded the treatment will end. If significant reduction in the size of the tumor is observed, a third and final cycle will be done.
* After the last cycle of chemotherapy is done, radiation therapy will be performed twice daily for 6-7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of squamous cell carcinoma of head and neck
* Patients will previously untreated stage III or IV squamous cell carcinoma.
* Patients with locally recurrent disease after surgery.
* Life expectancy of longer than 3 months.
* Kidney function: 1.5 or a 24 hour creatinine clearance of > 30ml/min
* Liver function: SGOT < 1.5 X upper normal limit and alkaline phosphatase of < 2.5 X upper normal limit.
* WBC greater than or equal to 4,000/mm
* Platelet count greater than or equal to 100,000/mm
* Hemoglobin greater than or equal to 10gm/dl
* Patients of child-bearing age must use effective methods of contraception.

Exclusion Criteria:

* Patients treated with previous chemotherapy or radiotherapy for head and neck cancer.
* Patients with concurrent malignancy of any site except limited basal cell carcinoma, squamous carcinoma of the skin or carcinoma in situ of the cervix.
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1997-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of taxotere, cisplatin, 5-fluorouracil and leucovorin.

SECONDARY OUTCOMES:
To evaluate the side effects of a four day outpatient regimen with taxotere, cisplatin, 5-fluorouracil and leucovorin
to obtain preliminary information about the effectiveness of the drug combination.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Colevas AD, Norris CM, Tishler RB, Lamb CC, Fried MP, Goguen LA, Gopal HV, Costello R, Read R, Adak S, Posner MR. Phase I/II trial of outpatient docetaxel, cisplatin, 5-fluorouracil, leucovorin (opTPFL) as induction for squamous cell carcinoma of the head and neck (SCCHN). Am J Clin Oncol. 2002 Apr;25(2):153-9. doi: 10.1097/00000421-200204000-00010. PMID 11943893
- [Background] Haddad R, Colevas AD, Tishler R, Busse P, Goguen L, Sullivan C, Norris CM, Lake-Willcutt B, Case MA, Costello R, Posner M. Docetaxel, cisplatin, and 5-fluorouracil-based induction chemotherapy in patients with locally advanced squamous cell carcinoma of the head and neck: the Dana Farber Cancer Institute experience. Cancer. 2003 Jan 15;97(2):412-8. doi: 10.1002/cncr.11063. PMID 12518365